CLINICAL TRIAL: NCT02982733
Title: Ankaferd Blood Stopper as a New Strategy to Avoid Early Complication After Transradial Coronary Angiography: A Randomized, Placebo-Controlled Clinical Trial
Brief Title: Ankaferd Blood Stopper for Hemostasis After Transradial Coronary Angiography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Sevket Gorgulu, Prof. Dr., Acibadem University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ATADEK2016/17-4
Record Dates: First submitted 2016-11-23; First posted 2016-12-05 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Radial Artery Injury; Hematoma; Bleed
MeSH Terms: conditions — Hematoma; Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ABS (Active Comparator): Ankaferd blood stopper
  Interventions: Other: ABS
- CS (Placebo Comparator): Conventional sterile gauze
  Interventions: Other: CS
- TR BAND (Active Comparator): Dedicated hemostatic device
  Interventions: Device: TR Band

INTERVENTIONS:
Other: ABS — Ankaferd Blood Stopper
  Arms: ABS
Device: TR Band — Transradial band
  Arms: TR BAND
Other: CS — Sterile Gauze
  Arms: CS

SUMMARY:
In 2008 Goker et al, introduced Ankaferd Blood Stopper (ABS) as a new hemostatic drug. Recently, ABS has been shown to produce local hemostasis by implementing topically after major arterial vessel injury. Reducing the compression time during patent hemostasis by facilitating hemostasis may decrease RAO. To test this hypothesis the investigators planned a three arm randomized study to evaluate the safety and efficacy of Ankaferd blood stopper in adjunct to short-time compression, compared to either short-time compression with conventional sterile gauzes or with a TR band after transradial diagnostic procedures.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients undergoing transradial elective diagnostic coronary procedures between November 2016 and November 2017 at the catheterization laboratory of Acibadem University Kocaeli Hospital were considered to be enrolled in the study.

Exclusion Criteria:

* The only exclusion criteria were an abnormal Barbeau's test before puncture and failure to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Radial artery occlusion assessed by reverse Barbeau's test | 24 hours

SECONDARY OUTCOMES:
Bleeding | 2 hours
  any kind of bleeding defined as ml after the removal of hemostatic dressings or devices
Hematoma | 24 hours
  hematomas larger then >5cm

CONTACTS AND LOCATIONS:
Overall Officials: Sevket Gorgulu, Prof, Study Chair — Acibadem University
Locations (1):
- Acibadem University, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Gorgulu S, Norgaz T, Sipahi I. Ankaferd blood stopper as a new strategy to avoid early complications after transradial procedures: A randomized clinical trial. J Interv Cardiol. 2018 Aug;31(4):511-517. doi: 10.1111/joic.12514. Epub 2018 Apr 17. PMID 29667233